CLINICAL TRIAL: NCT06979661
Title: Trial of ctDNA of Guidance to Determine PostOperative Radiation Therapy (PORT) for Minimal Residual Disease (MRD) for Lung Cancer: the MRD-PORT Trial
Brief Title: Trial of ctDNA of Guidance to Determine PostOperative Radiation Therapy
Acronym: PORT
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Salma Jabbour, MD, Professor of Radiation Oncology, Rutgers, The State University of New Jersey
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 032411
Record Dates: First submitted 2025-05-13; First posted 2025-05-20 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Lung Cancer; Non Small Cell Lung Cancer; Lung Cancer Recurrent
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single-Arm - ctDNA-Guided Treatment (Experimental): This single-group interventional arm evaluates the feasibility and impact of ctDNA testing in guiding adjuvant treatment decisions.
  Interventions: Diagnostic Test: Haystack™ ctDNA Assay

INTERVENTIONS:
Diagnostic Test: Haystack™ ctDNA Assay — A personalized, tumor-informed circulating tumor DNA (ctDNA) test that analyzes blood samples to detect minimal residual disease (MRD) and guide postoperative treatment decisions for patients with Stage II-III non-small cell lung cancer (NSCLC) following surgical resection. The test results will help determine whether patients should receive postoperative radiation therapy (PORT) and/or systemic therapy adjustments.

SUMMARY:
Primary Objective:

Evaluate the role of ctDNA positivity in decision making for postoperative therapy for non-small cell lung cancer. The plan for postoperative therapy will be declared after pathology report review and before the ctDNA result. We will assess if ctDNA result changed the planned therapy.

Secondary Objectives:

Evaluate personalized postoperative Chemo/ICPI/Targeted Therapies/Radiation Therapy in clearing ctDNA Evaluate the disease-free survival (DFS) and overall survival (OS) of stage II/III lung cancer patients with postoperative ctDNA positive status

Exploratory Objective:

Evaluate radiomics features based on serial CT thoracic CT scans to determine if radiomic features can be associated with ctDNA positivity/negativity.

DETAILED DESCRIPTION:
This is a pilot, single-arm interventional study evaluating the use of the Haystack™ circulating tumor DNA (ctDNA) assay to guide postoperative radiation therapy (PORT) and systemic therapy decisions for patients with Stage II-III non-small cell lung cancer (NSCLC) who have undergone surgical resection. The study aims to assess whether ctDNA monitoring can effectively detect minimal residual disease (MRD) and improve post-surgical treatment strategies.

ELIGIBILITY:
Inclusion Criteria:

1. Have provided signed informed consent for the trial
2. Aged ≥18 years at the time of informed consent
3. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
4. Diagnosed with histologically confirmed Stage II-III NSCLC and undergone surgical resection of lung tumor
5. No active second cancers/malignancy
6. Patients that received preoperative therapy (including chemotherapy and immunotherapy or others) are eligible
7. Willing and able to comply with all aspects of the protocol
8. Standard of care therapy and methods as per institution and investigator discretion -

Exclusion Criteria:

Exclusion Criteria

1. Discontinued treatment due to a Grade 3 or higher AEs with chemotherapy or immunotherapy or targeted therapy agent
2. With a history of another primary malignancy within the past 2 years that is considered an active malignancy by the enrolling physician.
3. Have known active CNS metastases and/or carcinomatous meningitis.
4. Have a history of (non-infectious) pneumonitis that required steroids or have current pneumonitis.
5. Have a history of interstitial lung disease.
6. Have a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the participant's participation for the full duration of the study, or is not in the best interest of the participant to participate, in the opinion of the treating investigator. -

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2028-06-01 (Estimated); Study Completion 2029-06-01 (Estimated)

PRIMARY OUTCOMES:
Detection of Circulating Tumor DNA (ctDNA) Post-Surgery | Baseline, 2-4 weeks, 3 months, 6 months, and 12 months post-surgery
  This outcome will assess the presence or absence of circulating tumor DNA (ctDNA) in blood samples collected at multiple time points following surgical resection of Stage II-III non-small cell lung cancer (NSCLC). The Haystack™ ctDNA assay will be used to detect minimal residual disease (MRD), and results will be evaluated for their ability to predict recurrence and guide postoperative radiation and systemic therapy decisions.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | Up to 3 years post-surgery
  This outcome measures the time from surgery to disease progression or recurrence, as determined by imaging, clinical assessment, or rising ctDNA levels detected via the Haystack™ ctDNA assay.
Overall Survival (OS) | Up to 5 years post-surgery
  The time from surgery to death from any cause. This will assess whether ctDNA-guided treatment impacts long-term survival outcomes in patients with Stage II-III NSCLC.
Change in ctDNA Levels Over Time | Baseline, 2-4 weeks, 3 months, 6 months, and 12 months post-surgery
  Measures the change in ctDNA levels detected in serial blood draws, evaluating whether fluctuations correlate with treatment response, recurrence risk, or progression.

CONTACTS AND LOCATIONS:
Locations (1):
- Rutgers Cancer Institute, New Brunswick, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No